CLINICAL TRIAL: NCT03285347
Title: The Effect of Computer-based Cognitive Training on Attention and Executive Functions in Patients With Parkinson's Disease
Brief Title: Effect of Computer-based Cognitive Training on Attention and Executive Functions in Patients With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Katrine Sværke, Stud. Psych., Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: H-17000220
Record Dates: First submitted 2017-09-14; First posted 2017-09-18 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Parkinson Disease; Executive Dysfunction
Keywords: parkinson; executive dysfunction; attention; computer-based cognitive training
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Two intervention Groups training with each their computer-based cognitive programme, one control Group receiving no intervention except for the same amount of follow-ups as the two intervention Groups.
Who Masked: Outcomes Assessor
Masking Description: Before and after the intervention period, the patients are tested in a neuropsychological battery to asses their executive functioning. The tester is blinded to the Group allocation of the patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Brain+ Evolution (Experimental): Intervention: Training with computer-based programme Brain+ Evolution for 8 weeks, receiving follow-ups every second week.
  Computer-based cognitive training.
  Interventions: Device: Computer-based cognitive training
- Scientific Brain Training PRO (Experimental): Intervention: Training with computer-based programme Scientific Brain Training PRO for 8 weeks, receiving follow-ups every second week.
  Computer-based cognitive training.
  Interventions: Device: Computer-based cognitive training
- Control group (No Intervention): This Group receives no intervention except for the same amount of follow-ups as the two training Groups. This is done to ensure that an effect of training is not aqtually due to the follow-up's with a professional.

INTERVENTIONS:
Device: Computer-based cognitive training — Computer-based cognitive programmes are computer programmes designed as games with the aim of training patients in certain cognitive domains.
  Arms: Brain+ Evolution; Scientific Brain Training PRO

SUMMARY:
The current study adresses the effect of two different computer-based cognitive trianing programmes on attention and executive functions in patients with Parkinson's disease.

DETAILED DESCRIPTION:
The current study adresses the effect of two different computer-based cognitive training programmes (Brain+ Evolution and Scientific Brain Training PRO) on attention and executive functions in patients with Parkinson's disease. The patients are assigned to one of three groups. Two training groups with each their programme, and a control Group. The training groups will train at home for 8 weeks with follow-ups every second week. The control group will not train at home, but will also receive a follow-up with computer-based stimuli (computerized Card game) every second week, to minimize the possibility that a possible effect is due to the follow-up's with a professional, and not due to the computer training at home.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Parkinson's disease AND
* Montreal cognitive assesment (MOCA)-score between 22-28
* Motorically cabable of using an iPad
* Not receiving antipsychotic medicine
* No comorbid diseases which might influence the level of executive functioning, for an example ADHD or acquired brain damage

Exclusion Criteria:

* People without Parkinson's disease
* Parkinson's patients not included in the above inclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2020-02-29 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
SDMT | 2 minutes
  Symbol digit modalities test, neuropsychological test of processing speed
PDQ-39 | 20 minutes
  Parkinson's disease questionnaire; daily functioning and well-being in Parkinson's disease

SECONDARY OUTCOMES:
HADS | 10 minutes
  Hospital anxiety and depression screening
Digit span | 10 minutes
  Digit span Wais-IV; Working memory
Verbal fluency | 3 minutes
  S-Words, animal-names and A/F-words
Stroop colour/word test | 3 minutes
  Stroop colour/Word test, respone inhibition
Trail Making A and B | 5 minutes
  Trail Making A and B, cognitive flexibility

CONTACTS AND LOCATIONS:
Overall Officials: Annemette Løkkegaard, Ph.d., Study Director — Doctor
Locations (1):
- Bispebjerg Hospital, Copenhagen, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Svaerke K, Faerk AK, Riis A, Stiegnitz von Ehrenfels SEM, Mogensen J, Lokkegaard A. Effects of Computer-Based Cognitive Rehabilitation on Attention, Executive Functions, and Quality of Life in Patients with Parkinson's Disease: A Randomized, Controlled, Single-Blinded Pilot Study. Dement Geriatr Cogn Disord. 2021;50(6):519-528. doi: 10.1159/000520591. Epub 2022 Jan 5. PMID 34986487